CLINICAL TRIAL: NCT05877989
Title: Evaluation of Effectiveness of Combining High Protein Intake With Early Physical Exercise During Critical Illness to Maintain Muscle Mass in Intensive Care Unite Patient.
Brief Title: Evaluation of Effectiveness of Combining High Protein Intake With Early Physical Exercise During Critical Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Badr Eldin, Doctor Asmaa Badr Eldin, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34750/6/21
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Amino Acids; Exercise

STUDY DESIGN:
Intervention Model Description: Patients will receive the amino acid intervention that is provided in addition to 'usual care' enteral and/or parenteral nutrition either enteral or parenteral to target a total protein delivery of 2.0g/kg/day. The physical exercise intervention will be delivered by trained nursing staff,and started as close to the time of randomisation as feasible (ie, within 24hours of randomization). The intervention group will receive exercise sessions, for up to 20 min duration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Patients will receive usual care in Intensive Care Unit (prescription of a standard nutrition formula (at approximately 20 -25 kcal/ kg/day and protein intake 1.2 g/kg/day) once patients are hemodynamically stable.
  Interventions: Drug: Amino Acid
- Protein and exercise group (Active Comparator): patients will receive the amino acid intervention that is provided in addition to 'usual care' enteral and/or parenteral nutrition either enteral or parenteral to target a total protein delivery of 2.0g/kg/day. The physical exercise intervention will be delivered by trained nursing staff, and started as close to the time of randomization as feasible (within 24hours of randomization). The intervention group will receive exercise sessions, for up to 20 min duration (as tolerated by patient). The implementation of physical exercise intervention will be protocolized to provide passive exercise early before weaning and shift to active exercise after weaning and also graduated resistance during each session and between daily sessions.
  Interventions: Drug: Amino Acid; Procedure: Physical exercise

INTERVENTIONS:
Drug: Amino Acid — Amino acid enteral and/or parenteral nutrition either enteral or parenteral to target a total protein delivery of 2.0g/kg/day.
Procedure: Physical exercise — The physical exercise intervention will be delivered by trained nursing staff, and started as close to the time of randomization as feasible (within 24hours of randomization). The intervention group will receive exercise sessions, for up to 20 min duration (as tolerated by patient).The implementation of physical exercise intervention will be protocolized to provide passive exercise early before weaning and shift to active exercise after weaning and also graduated resistance during each session and between daily sessions.
  Arms: Protein and exercise group

SUMMARY:
Assessment of Effectiveness of combined high protein intake with early physical exercise by ultrasound measurement of rectus femoris muscle thickness in Intensive Care Unite mechanically ventilated patients.

DETAILED DESCRIPTION:
Muscle wasting and weakness is a frequent finding in critically ill patients and is associated with worse short- and long-term outcomes like delayed liberation from mechanical ventilation, longer Intensive Care Unit and hospital stay, worse physical function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients in age group 18-60 years
* Expected Intensive Care Unit stay >4days after enrolment (to permit adequate exposure to the proposed intervention)
* Previously healthy, Well-nourished, subjects (nutric score=0)

Exclusion Criteria:

* Renal, liver or heart disease or chronic obstructive pulmonary disease
* Previous immune abnormalities (including treatment with corticosteroids)
* Past history of nutritional problems, chronic use of drugs (as drugs inducing myopathies) or orthopedic problems (such as skeletal fractures or immobilization) in the previous 2 years
* Neuromuscular diseases and patients with amputated lower limbs
* Past or recent history of cancer
* Long term critically ill patients shifted from other hospitals
* Pregnant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Quantitative changes (cross-section diameter) of rectus femoris muscle | Up to 30 days of Surgical Intensive Care Unit stay.
  Rectus femoris cross-sectional area (RFCSA) will be measured by B-mode ultrasonography using a 3 to 12 MHz transducer array. Patient will be positioned supine in 30° upper body elevation, with legs extended and muscles relaxed. The point that represented 60% of the distance from the anterior superior iliac spine to the superior border of the patella will be identified. The ultrasound probe will be positioned perpendicularly along the superior aspect of the right thigh and transverse images of the rectus femoris will be obtained. A copious amount of gel will be applied to minimize tissue compression. The inner echogenic line of the Rectus Femoris will be traced manually on a frozen image and RFCSA will be calculated by planimetric technique.

SECONDARY OUTCOMES:
Functional capacity. | Up to 30 days of Surgical Intensive Care Unit stay.
  Ultrasound evaluation of the rectus femoris muscle
Duration of mechanical ventilation. | Up to 30 days of Surgical Intensive Care Unit stay.
  Duration of mechanical ventilation.
Length of Surgical Intensive Care Unit stay. | Up to 30 days
  Length of Surgical Intensive Care Unit stay.
Mortality rate in Surgical Intensive Care Unit | Up to 30 days
  Rate of death in Surgical Intensive Care Unit
Rate of hospital acquired infection. | Up to 30 days
  Rate of hospital acquired infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author for one year after study completion.
Supporting Information: Study Protocol